CLINICAL TRIAL: NCT02237755
Title: Prospective Randomized Trial on the Effect of Clomiphene Citrate Administration in Women With Poor Ovarian Reserve Undergoing Controlled Ovarian Stimulation for IVF. Impact on Stimulation Characteristics and Pregnancy Outcome.
Brief Title: Clomiphene Citrate in Combination With Gonadotropins for Ovarian Stimulation in Women With Poor Ovarian Response.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Athens (Other)
Collaborators: Lito Maternity Hospital (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, Associate Professor of Obstetrics and Gynecology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NV25042014
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Female Infertility
Keywords: Clomiphene citrate; IVF; Pregnancy Rates; Ovarian Reserve
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene; Gonadotropins; Menotropins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomiphene citrate (Active Comparator): Administration of Clomiphene citrate in combination with gonadotropins according to a short stimulation GnRH antagonists protocol.
  Interventions: Drug: Clomiphene citrate; Drug: Gonadotropins
- Gonadotropins (Active Comparator): Patients in this group will be stimulated according to a short stimulation protocol with gonadotropins and GnRH antagonists.
  Interventions: Drug: Clomiphene citrate; Drug: Gonadotropins

INTERVENTIONS:
Drug: Clomiphene citrate — clomiphene citrate 100mg/day will be added to the standard gonadotropin regiment
  Other Names: Clomiphene citrate 50 mg/tab; Cerpafar 50 mg/tab
Drug: Gonadotropins — All patients will be stimulated with a fixed GnRH-antagonist protocol. Ovarian stimulation will be initiated with 450 IU of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH.
  Other Names: Menopur 75IU , Gonal

SUMMARY:
Coadministration of various drugs used for ovarian stimulation can increase the efficiency of IVF especially in poor responders. The investigators hypothesize that ovarian response of those patients could improve by using combination of clomiphene citrate with gonadotropins in infertile women with poor response to gonadotrophin administration only.

DETAILED DESCRIPTION:
Patients diagnosed with poor ovarian response will be included in the study. The definition of poor response was based on the presence of at least one of the following criteria: Age > 40 years old, day 2 FSH >9.5 mIU/ml, AMH < 2ng/ml ,at least one previous COH with less than 3 oocytes retrieved, at least one cancelled attempt due to poor response, estradiol less than 500 pg/ml on the day of HCG. All patients will be counseled regarding their prognosis and other treatment options including oocyte donation as well as adoption were also presented and discussed in detail. Early follicular phase FSH, estradiol (E2) and Anti-Mullerian Hormone (AMH) will be measured prior to the initiation of treatment. Women in the Clomiphene group will receive 100-150 mg of Clomiphene citrate once per day for 5 days in combination with gonadotropins according to short GnRH-antagonist protocol: all women will have measurements of serum FSH and estradiol and a pelvic sonogram on the second day of their cycle. Providing that serum FSH is < 17 mIU/ml and estradiol is < 70 pg/ml on day 2 , ovarian stimulation will be initiated with 100-150 mg of Clomiphene citrate in combination with 450 IU of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH. All patients will be re-evaluated on day 5 of the stimulation, and dosage adjustments will be made and the antagonists (Cetrorelix or ganirelix 0.25 mg/day) will be initiated. When at least 2 follicles reach an average diameter of 17 mm, final oocyte maturation will be triggered with 10,000IU of hCG ( Pregnyl, Organon, Greece Inc.). Oocyte retrieval will be performed 34 to 36 hours later. All patients will undergo ICSI. Patients with successful fertilization will have embryo transfer under sonographic guidance on day 3 after retrieval. Women in the Gonadotropin group will receive only gonadotropins according to short GnRH-antagonist protocol as it was mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Women with poor response to ovarian stimulation. The definition of poor response was based on the presence of at least one of the following criteria: Age > 40 years old, day 2 FSH >9.5 mIU/ml, AMH < 2ng/ml ,at least one previous COH with less than 3 oocytes retrieved, at least one cancelled attempt due to poor response, estradiol less than 500 pg/ml on the day of HCG.

Exclusion Criteria:

* All other women that do not fulfill the above mentioned criteria

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | 14 days after embryo transfer
  At the completion of the ovarian stimulation patients that will proceed to transfer and have a positive pregnancy test will have sonographic evaluation for confirmation of clinical pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Vlahos, Assoc. Prof., Study Chair — University of Athens, 2nd Department of Obstetrics and Gynecology; Olga Triantafyllidou, MD, Principal Investigator — University of Athens School of Medicine